CLINICAL TRIAL: NCT05428683
Title: Assistant Professor, Ophthalmology Department, Al Azhar University
Brief Title: Intravitreal Triamcinolone and Moxifloxacin Injection After Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emad Abdel Aal Saliem (Other)
Responsible Party: Sponsor-Investigator, Emad Abdel Aal Saliem, Assistant professor, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1221975
Record Dates: First submitted 2022-03-18; First posted 2022-06-23 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Pharmacological Action
Keywords: Endophthalmitis
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Intervention Model Description: cataract surgery followed by intravitreal injection of triamcinolone and moxifloxacin combination as a prophylaxis against endophthalmitis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prophylactic measures against post-operative inflammations (Other): Usage of triamcinolone and moxifloxacin combination to be injected intravitreally by using 30 G needle.
  Interventions: Drug: intra-vitreal triamcinolone-moxifloxacin injection after cataract surgery as a prophylactic measures against post-operative endophthalmitis

INTERVENTIONS:
Drug: intra-vitreal triamcinolone-moxifloxacin injection after cataract surgery as a prophylactic measures against post-operative endophthalmitis — At the end of surgery, 4mg triamcinolone acetonide and 0.2mg moxifloxacin from 0.5 moxifloxacin preservative-free eye drop) were injected once inferotemporally 3.5 mm posterior to the limbus via pars plana into the vitreous cavity by using 30 G needle.

SUMMARY:
This study aims to evaluate the short-term effects and safety of prophylactic intra-vitreal injection of triamcinolone-moxifloxacin combination after cataract surgery. 84 patients underwent cataract surgery associated with intra-vitreal injection of triamcinolone-moxifloxacin combination after surgery.

DETAILED DESCRIPTION:
All the patients underwent the surgical removal of cataract by the same surgeon according to the standard protocols for modern phacoemulsification. Surgery was done under local anesthesia by peri-bulbar injection of local anesthetic. All operations were performed in an operating room by using an operating microscope under complete aseptic condition by using 10% povidone iodine solution applied to the skin of eye lid, eye lashes, side of the nose, eye brow and the skin of forehead. Before the operation, sterile drape and eyelid speculum were used, then 5% povidone iodine solution was applied to the bulbar conjunctiva and fornices for about 5 minutes, then was irrigated by balanced salt solution (BSS).

All the patients were followed up at the 1st day, 1st week, 1st month and at the 3rd month after the operation. At each visit the followings should be assessed: the post-operative refraction, the best corrected visual acuity and anterior and posterior segments examination for any sign of postoperative inflammation as cells and flare. Intra-ocular pressure (IOP) assessment and optical coherence tomography (OCT) images were also taken at the 1st and the 3rd postoperative months to assess the central macular thickness in suspected cases of cystoid macular edema (CME) based upon symptoms or signs observed on fundus examination, were confirmed by OCT of the macula through subjective interpretation via presence of cysts or an objective measurement of retinal thickness > 250 microns.

ELIGIBILITY:
Inclusion criteria: Patients underwent uncomplicated cataract surgery with:

* A significant cataract.
* Good control of diabetes mellitus (DM) and hypertension (HPT) if present.
* Visual acuity not less than hand movement (HM).

Exclusion criteria:

The followings were the exclusion criteria:

* The use of systemic or topical steroids, topical ophthalmic antibiotics, or non-steroidal anti-inflammatory drugs (NSAIDs) for one week before operation.
* Make an additional procedure at the same time with cataract surgery.
* Those with uncontrolled glaucoma or with marked visual field defect .
* Those with a significant macular edema due to DM, HPT, retinal vein occlusion (CRVO) or due to any previous inflammatory condition.
* Those with blepharitis or any other local disease interfering with surgical intervention or affecting on the surgical outcome.
* Occurrence of intraoperative complications as posterior capsular rupture or postoperative complications as retained lens fragment.

Ages: 48 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Post operative best corrected visual acuity | at the end of 3rd month.
  describe the differences between pre & post operative best corrected visual acuity by snellen's chart. The mean BCVA showed a statistically significant differences between the preoperative and the postoperative values, where the main BCVA improved from 1.21±0.27 logMAR before operation (at baseline) to 0.19±0.14 logMAR at the 3rd month. For statistical analysis, the best- corrected visual acuity data were transformed to LogMAR. Investigators calculated the mean, standard deviation, range, confidence interval, and Pearson correlation.
A condition of the eye after cataract surgery without use of topical medications. | purpose of this study is to evaluate the efficacy of these used drugs after surgery not before it during follow up period at the end of 3rd month.
  By SLITLAMP examination, investigators search for signs of postoperative endophthalmitis or inflammations as cells or flare that required supplemental anti-inflammatory medications. So, evaluate the use of triamcinolone-moxifloxacin combination after cataract surgery when injected intra-vitreally against postoperative endophthalmitis and/or other intraocular inflammations without use of topical anti-infective and/or anti-inflammatory medications whether before or even after cataract surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Emad A Saliem, Study Director — Assistant Prof of ophthalmology, Al Azhar university
Locations (1):
- Emad AbdelAal Saliem, Ţahţā, Sohag Governorate, Egypt